CLINICAL TRIAL: NCT01206699
Title: Involvement of Transverso-sacral- Neo- Articulations or of Transverso-iliac Articulations in Chronic Lumbago: Prospective Multicentric , Double-Blinded, Randomized of the Efficacy of corticoïd Infiltration Versus Physiological Solution Infiltration
Brief Title: Involvement of Transverso-sacral- Neo- Articulations or of Transverso-iliac Articulations in Chronic Lumbago
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: after 4 years of recruitment only 16 patients have been included. Due to this low rate of recruitment it was decided to stop the study
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10/3-N
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2010-09

CONDITIONS: Subjects Suffering of Lateralized Lumbago on Side of the Malformation (Neo-articulation)
MeSH Terms: interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- corticoid (Experimental): Active arm : anesthetic bloc (1 ml of lidocaïne 1%) immediately followed with corticoid (altim® 1.5 ml)
  Interventions: Drug: corticoid (altim® 1.5 ml)
- physiological solution (Placebo Comparator): Control arm: anesthetic bloc (1 ml of lidocaïne 1%) immediately followed with physiological solution (1.5 ml)
  Interventions: Drug: physiological solution (1.5 ml)

INTERVENTIONS:
Drug: corticoid (altim® 1.5 ml) — Active arm : anesthetic bloc (1 ml of lidocaïne 1%) immediately followed with corticoid (altim® 1.5 ml)
  Arms: corticoid
Drug: physiological solution (1.5 ml) — Control arm: anesthetic bloc (1 ml of lidocaïne 1%) immediately followed with physiological solution (1.5 ml)
  Arms: physiological solution

SUMMARY:
The specific aim of this study is to determine whether, when treated with corticoid infiltration, certain chronic lumbagos could be explained by the presence of a neo-articulation.The primary criteria is to determine the difference between the mean pain during the latest 24 hours preceding the infiltration and the mean pain preceding the visit S4 (visit 4 weeks after the infiltration)

ELIGIBILITY:
Inclusion Criteria:

* Adult with age equal or above to 18.
* Subject affiliated to French health insurance (Sécurité Sociale)
* Lateralized lumbago on side of the neo-articulation evolving since more than 3 months
* Mechanical pain, lumbar low level or gluteal without sciatic irradiation (pain above the knee)
* Mean pain during the latest 24 hours above 4 on an analogic visual scale (from 0 to 10)- Pain induced by palpation in regards to the neo-articulation
* Pain not relieved by medical treatment with non steroids anti- inflammatory drugs or antalgics
* No clinical proof for a discal origin : inducing factor, impulsiveness, spinal syndrome, true Lasègue
* transverse-sacral abnormality of IIb, IIIa, IIIc or IV type with neo-articulation lateralized on side of pain
* Informed consent form signed

Exclusion Criteria:

* Age below 18
* Clinical arguments in favour of a discal origin
* Pregnant women or women that could become pregnant the day of the infiltration
* Diabetic patient
* Patient unable to understand the protocol
* No autonomy for coming to the hospital (no budget allocated for patient transportation)
* Hypersensitivity to local anesthetics with "liaison amide"
* Hypersensitivity to one of the components
* Porphyria- Local or generalized infection, suspiscion of infection
* Severe troubles of coagulation, anti-coagulant treatment taken
* Bilateral lumbago with bilateral neo-articulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
To determine the difference between the mean pain during the latest 24 hours preceding the infiltration and the mean pain preceding the visit S4 (visit 4 weeks after the infiltration) | week 4
  To determine whether, when treated with corticoid infiltration, certain chronic lumbagos could be explained by the presence of a neo-articulation.The primary criteria is to determine the difference between the mean pain during the latest 24 hours preceding the infiltration and the mean pain preceding the visit S4 (visit 4 weeks after the infiltration)

SECONDARY OUTCOMES:
To determine whether the improvement by the infiltration of corticoid is present at visit J7 (visit 7 days after the infiltration) and at visit S12 (visit 12 weeks after the infiltration)
To determine whether an anesthetic positif bloc (decrease of the pain of more than 75 % during the hour that follows the infiltration) is a predictive factor of the final result
To determine whether corticoïd infiltration can decrease the intake of drugs et decrease the functional handicap

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hospital of La Roche/Yon, La Roche/Yon
  - Nantes Hospital, Nantes